CLINICAL TRIAL: NCT02412852
Title: A Randomized, Double-blinded, Phase 2a Study to Assess the Safety and Pharmacokinetics of a Sustained Release Formulation of Sodium Nitrite (TV1001sr) in Patients With Diabetic Neuropathic Pain (DNP)
Brief Title: A Phase 2a Study to Assess Safety & Pharmacokinetics of Sustained Release Sodium Nitrite in Patients With Diabetic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TheraVasc Inc. (Industry)
Collaborators: Kettering Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TheraVasc-TV1001-003
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Diabetes
Keywords: neuropathy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): One placebo tablet administered twice daily for 12 weeks.
  Interventions: Drug: Placebo
- 40 mg TV1001sr (Active Comparator): One 40 mg enteric coated sustained release, sodium nitrite tablets administered twice daily.
  Interventions: Drug: Sodium nitrite
- Placebo (2) (Placebo Comparator): Two placebo tablets administered twice daily for 12 weeks.
  Interventions: Drug: Placebo
- 80 mg TV1001sr (Active Comparator): Two 40 mg enteric coated sustained release, sodium nitrite tablets administered twice daily.
  Interventions: Drug: Sodium nitrite

INTERVENTIONS:
Drug: Sodium nitrite — Sustained release formulation of sodium nitrite
  Other Names: TV1001sr
  Arms: 40 mg TV1001sr; 80 mg TV1001sr
Drug: Placebo — Placebo tablets containing same excipients and coatings used in the active tablets, without sodium nitrite being added.
  Arms: Placebo; Placebo (2)

SUMMARY:
In this study, subjects with diabetic neuropathic pain (DNP) will be treated for 12 weeks with either placebo, 40 or 80 mg sustained release sodium nitrite (TV1001sr) twice daily. Primary endpoints will be safety and pharmacokinetics. Assessment of the study medications affects on pain following treatment will also be recorded.

DETAILED DESCRIPTION:
This is a dose-ranging study to evaluate the safety, pharmacokinetics, and tolerability of multiple doses of an oral, sustained release formulation of sodium nitrite (TV1001sr) in subjects with DNP. The primary objective is to assess the safety and tolerability of multiple doses of twice daily 40 mg and 80 mg TV1001sr compared with placebo over a 12 week treatment period and the pharmacokinetics of the sustained release formulation of sodium nitrite. Secondary objectives are to evaluate the pharmacokinetics and markers of functional improvement including pain questionnaires, quantitative sensory testing and changes in markers of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects must be post-menopausal, sterilized or using suitable birth control
* Diagnosis of diabetes (HbA1c > 6.0)
* Diagnosis of diabetic peripheral neuropathy pain in feet
* Presence of ongoing diabetic neuropathic for at least 3 months
* A pain score of greater than or equal to 4 on the Numerical Pain Rating Scale at screening
* Ability to provide written informed consent

Exclusion Criteria:

* Patients with fibromyalgia or regional pain caused by lumbar or cervical compression
* History or diagnosis of significant neurological disease
* History and diagnosis of clinically significant psychiatric diseases
* Serious liver disease
* Poorly controlled diabetes
* Hypersensitivity to sodium nitrite or related compounds
* Life expectancy < 6 months
* A chronic illness that may increase the risks associated with this study
* Active malignancy requiring active anti-neoplastic therapy that will, in the opinion of the investigator, interfere with study treatment or participation
* Pregnant or nursing women
* Current diagnosis of alcohol or other substance abuse
* Current use of sildenafil or other phosphodiesterase Type 5 Inhibitors
* History of methemoglobinemia, (met-Hb ≥ 15%)
* Subject is involved in litigation or receives worker's compensation
* Inability to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04-28 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2017-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amol Soin, PhD, Principal Investigator — Ohio Pain Clinic
Locations (1):
- Ohio Pain Clinic, Centerville, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to the PI of the trial, summary information will be published and shared with other researchers.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: One placebo tablet administered twice daily for 12 weeks.
  Placebo: Placebo tablets
- Placebo (2): Two placebo tablets administered twice daily for 12 weeks.
  Placebo: Placebo tablets
Period: Overall Study
Arm/Group | Placebo | 40 mg TV1001sr | Placebo (2) | 80 mg TV1001sr
Started | 4 | 8 | 5 | 9
Completed | 4 | 7 | 5 | 8
Not Completed | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 40 mg TV1001sr | Placebo (2) | 80 mg TV1001sr | Total
Number analyzed (Participants) | 4 | 8 | 5 | 9 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 2 | 7 | 16
  >=65 years | 3 | 2 | 3 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 4 | 5 | 12
  Male | 4 | 5 | 1 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 8 | 5 | 9 | 26
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 5 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Reporting of Adverse Events During 12 Week Study Period
Description: The primary objective of this clinical study is to evaluate the safety and tolerability of multiple doses of twice daily 40mg and 80mg sustained release sodium nitrite compared with placebo over a 12 week treatment period. The following safety parameters will also be assessed: concomitant medication usage, physical examination, vital signs, Comprehensive Metabolic Panel, and complete blood count. Assessment of acute adverse events (i.e., drop in blood pressure, dizziness) after administration of each dose level. Counts are number of subjects reporting at least 1 Adverse Event. The total Adverse Events recorded in each cohort is also reported.
Time Frame: 12 weeks
Population: Randomized population including dropouts.
Measure: Number; unit: Adverse Events
Groups:
- Combined Placebo: A combination of the once/day and twice/day placebo groups.
- 40 mg TV1001sr: Treatment twice daily with 40 mg sustained release sodium nitrite
- 80 mg TV1001sr: Treatment with 80 mg (2 x 40 mg tablets) twice daily with sustained release sodium nitrite
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 8 | 9
Adverse Events
  Subjects reporting at least one Adverse Event | 9 | 8 | 7
  Total Adverse Events reported in each cohort | 29 | 23 | 24

2. Secondary Outcome: Pharmacokinetics (Blood Levels of Nitrite)
Description: Blood levels of nitrite will be assessed for 6 hours post-administration on the initial dosing visit.
Time Frame: 1 day
Population: All subjects who were randomized.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 8 | 9
ng/ml | 1399 (47) | 9699 (10199) | 9905 (12383)
Statistical Analysis 1: Comparison: Combined Placebo vs 40 mg TV1001sr vs 80 mg TV1001sr; Test type: Other; ]The pharmacokinetics data are particularly sparse, and therefore substantial interpolations and imputations were required to produce an analyzable data set. Consequently, while not ideal, the Last Observation Carried Forward method was used for these data. There was a large amount of missing data which required imputation to determine results. The large amount of interpolations and imputations required for the pharmacokinetic analysis means that the pharmacokinetic results will need to be interpreted with caution. 3 X 3 Analysis of Variance used to compare Placebo to the two active groups. Missing data required imputation of available data

3. Secondary Outcome: The Number of Participants Who Reported Use of Analgesic or Medications for Neuropathic Pain.
Description: Daily patient reported use of analgesic or medications for neuropathic pain. The use of medications were recorded at the baseline visit and during both the intermediate and final visit for each subject. All subjects used at least one prescription pain medication, other than one subject in the 80-mg dose cohort who used only ibuprofen to control pain. Most subjects used more than one prescription pain medication. There was no change in use of pain medications during the trial period.
Time Frame: 12 weeks
Population: Analyzed only those subjects who completed 12 weeks of testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 7 | 8
Participants
  Subjects using any medicine to treat pain | 9 | 7 | 8
  Subjects using Gabapentin | 6 | 6 | 3
  Subjects using Lyrica | 4 | 4 | 4
  Subjects using Morphine | 2 | 1 | 0
  Subjects using Tramadol | 1 | 3 | 3
  Subjects using Cymbalta | 1 | 1 | 2
  Subjects using Flexeril | 1 | 0 | 2
  Subjects using Naproxen | 1 | 3 | 0
  Subjects using Percocet | 3 | 1 | 0
  Subjects using Vicodin | 2 | 2 | 1

4. Secondary Outcome: Assessment of Patients Reported Pain Through Composite Analysis of Pain Questionaires.
Description: Subjects completed the Brief pain inventory (BPI), RAND 36 questionnaire, neuropathic pain symptom inventory (NPSI) and Short Form McGill Pain Questionnaire at each visit for these self-reported questionnaires. The BPI is a questionnaire that measures the patient's subjective perception of pain, its exacerbating and alleviating factors, and perceived effect on functional status; the NPSI is a questionnaire that measures the symptoms associated with neuropathic pain; the Short Form McGill Questionnaire subjectively assesses the patients perception of pain described by commonly used adjectives associated with pain. NPSI is average of 12 questions, range from 0 (no pain) to 120 (maximal pain); For BPI severity and interference, questions are scored from 0-10, then there average score for each subsection is calculated (the higher the score, the worse the response); Scores on McGill range from 0-10, lower associated for less pain, then averaged for each sub score and total score.
Time Frame: Baseline (visit 1) and 12 weeks (visit 3)
Population: NPS is a sum of total scores, McGill and BPI an average of the scores for each question.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 7 | 8
units on a scale
  NPSI: Total-V1 | 47.4 [7 to 75] | 34.7 [18 to 80] | 56.0 [21 to 83]
  NPSI: Total-V3 | 43.4 [9 to 81] | 30.0 [0 to 76] | 46.0 [6 to 73]
  BPI: Severity Score-V1 | 5.1 [1.25 to 7.5] | 4.3 [1.25 to 8.5] | 5.9 [2.5 to 9.3]
  BPI: Severity Score-V3 | 4.8 [1.5 to 7.8] | 3.8 [0.8 to 8.8] | 5.1 [2.0 to 8.3]
  BPI: Interferrence-V1 | 5.0 [0.0 to 9.7] | 4.4 [0.7 to 7.9] | 6.4 [2.0 to 8.5]
  BPI: Interferrence-V3 | 4.3 [0.0 to 10.0] | 4.2 [1.1 to 8.6] | 5.7 [3.1 to 8.9]
  McGill: Total-V1 | 5.1 [1.1 to 9.1] | 3.9 [1.8 to 7.6] | 4.8 [1.7 to 7.9]
  McGill: Total-V3 | 3.6 [0.4 to 7.5] | 2.5 [0.5 to 7.2] | 4.6 [0.5 to 7.0]
  McGill: Continuous-V1 | 5.0 [1.0 to 9.0] | 3.7 [0.9 to 7.2] | 4.4 [0.5 to 8.0]
  McGill: Continuous-V3 | 3.2 [0.0 to 6.6] | 1.9 [0.0 to 5.8] | 4.3 [0.7 to 7.5]
  McGill: Intermittent-V1 | 6.0 [0.0 to 9.7] | 4.6 [2.3 to 8.5] | 5.9 [0.3 to 8.0]
  McGill: Intermittent-V3 | 4.1 [0.0 to 9.2] | 2.8 [0.0 to 8.3] | 5.3 [0.0 to 7.3]
Statistical Analysis 1: Comparison: Combined Placebo vs 40 mg TV1001sr vs 80 mg TV1001sr; Test type: Other — ANOVA on only those subjects who completed testing; p = 0.05, ANOVA — The results were analyzed using an ANOVA with one between-subjects factor (Group: both placebo groups combined, 40 mg TV1001sr, and 80 mg TV1001sr); and one within-subjects factor (Visit: Visit 1, Visit 2, and Visit 3); The means of the three groups were further analyzed using a post hoc comparison procedure (the Scheffé test)

5. Secondary Outcome: Clinical Assessment of Pain. (Quantitative Sensory Testing)
Description: Quantitative sensory testing (QST) was conducted at each visit to determine patients sensitivity to pain. QST was assessed using a quantitative nerve conductance machine where nerves in the distal extremity are subjected to electrical stimulation to determine the sensory threshold of the skin. Nerve conductance measures how fast an electrical impulse moves through the nerve, and nerve velocity measures the speed at which an electrical impulse moves down a neuronal pathway.
Time Frame: 12 weeks
Population: Analyzed only the subjects that completed testing.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 7 | 8
meters per second
  Nerve Conductance: Baseline | 3.9 (1.4) | 3.4 (0.7) | 6.0 (2.9)
  Nerve Conductance: V2 | 4.3 (1.8) | 3.1 (0.9) | 5.2 (3.0)
  Nerve Conductance: V3 | 3.5 (1.2) | 3.2 (0.6) | 4.2 (1.5)
  Nerve Velocity: Baseline | 44.7 (6.5) | 41.1 (4.3) | 39.4 (8.2)
  Nerve Velocity: V2 | 40.1 (5.3) | 39.3 (7.8) | 42.3 (10.7)
  Nerve Velocity: V3 | 43.2 (6.4) | 37.7 (3.2) | 46.8 (4.2)
Statistical Analysis 1: Comparison: Combined Placebo vs 40 mg TV1001sr vs 80 mg TV1001sr; Test type: Other — The composite conduction measure and the composite velocity measure were analyzed using an Analysis of Variance with one between-subjects factor (Group: combined placebo, 40 mg TV1001, and 80 mg TV1001); and one within-subjects factor (Visit: Visit 1, Visit 2, and Visit 3); p = .15, ANOVA

6. Secondary Outcome: Assessment of Diabetes. (HbA1C Levels)
Description: HbA1C levels will be monitored at each visit to determine whether treatment reduces circulating glucose levels.
Time Frame: 12 weeks
Population: HbA1c blood levels were analyzed at baseline, V2 and V3
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 7 | 8
percentage of glycosylated hemoglobin
  Baseline | 7.7 (1.4) | 7.7 (1.2) | 8.5 (2.4)
  V2 | 7.3 (1.2) | 7.4 (0.9) | 7.9 (1.8)
  V3 | 7.6 (2.0) | 7.7 (1.6) | 8.2 (1.2)
Statistical Analysis 1: Comparison: Combined Placebo vs 40 mg TV1001sr vs 80 mg TV1001sr; Test type: Other — A 3 by 3 Analysis of Variance with one between-subjects factor (Combined placebo, 40 mg TV1001, or 80 mg TV1001) and one within-subjects factor (Visit 1, Visit 2, or Visit 3) was performed for HbA1c values; p = .36, ANOVA

7. Secondary Outcome: Assessment of Blood Oxygenation. (Pulse Oximetry)
Description: Pulse oximetry will be used at each visit to determine whether treatment improves oxygen levels in the blood.
Time Frame: 12 weeks
Population: Oxygen saturation was measured at baseline, V2 and V3.
Measure: Mean (Standard Deviation); unit: % Oxygenation
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
Number analyzed (Participants) | 9 | 7 | 8
% Oxygenation
  Baseline | 95.7 (2.6) | 95.6 (2.3) | 96.3 (1.7)
  V2 | 96.0 (3.0) | 96.4 (2.2) | 95.3 (3.2)
  V3 | 94.2 (2.8) | 96.0 (2.4) | 95.1 (2.4)
Statistical Analysis 1: Comparison: Combined Placebo vs 40 mg TV1001sr vs 80 mg TV1001sr; Test type: Other — ANOVA to compare differences from baseline to completion of testing; p = .93, ANOVA

ADVERSE EVENTS:
Time Frame: 9 months
Description: Asked subjects at each phone call and visit to report any adverse event.
Arm/Group | Combined Placebo | 40 mg TV1001sr | 80 mg TV1001sr
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 2/9 | 2/8 | 2/8
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Placebo (N=9) | 40 mg TV1001sr (N=8) | 80 mg TV1001sr (N=8)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pains (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile illness (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Placebo (N=9) | 40 mg TV1001sr (N=8) | 80 mg TV1001sr (N=9)
Headaches (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Urinary Disorders (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
Ulcers (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Swelling (General disorders) | 4 (4) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Numbness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No